CLINICAL TRIAL: NCT07233928
Title: Breast Cancer Organelle Properties and Protein Expression Atlas in the Three Immunohistochemical Subtypes of Breast Cancers
Acronym: ESPRESSOBREAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 25SEIN08
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Early Breast Cancer; Metastatic Breast Cancer
Keywords: breast cancer; organelle; lipid droplets; protein expression atlas and heterogeneity; metabolism
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The participants will be divided in 4 cohorts depending on the type of breast cancer (early stage [eBC] v. de novo metastatic [dnMBC]) and depending on the immunohistochemical subtype (triple negative, HER2+, luminal). The 4 cohorts will enroll independantly (in parallel).
  However, the sample collection schedule will differ depending on the treatment strategy. Three main treatment strategies have been identified:
  * Cohorts A, B and C (=early BC): with indication of neo-adjuvant treament
  * Cohorts A, B and C (=early BC): without indication of neo-adjuvant treatment
  * Cohort D (=dnMBC): metastatic treatment (with surgery if applicable)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early breast cancer (triple negative, HER2+, luminal) with indication of neo-adjuvant treatment (Other): * The following samples will be collected during the study :
    * Tumor sample (primitive tumor ± metastatic axillary lymph node) at: baseline, surgery, 1st recurrence
    * Blood samples at: baseline, mid-course of neo-adjuvant treatment, before and after surgery, end of systemic adjuvant treatment, every 6 or 12 months until the 1st recurrence or during 5 year follow-up period, following progressions/recurrences
    * Ascite and pleural fluid (when a puncture procedure is performed for clinical purposes) at: 1st recurrence, following progressions/recurrences
  * Data collection will be performed at baseline and then at each time point planned in the center for clinical standard of care assessment or clinical trial until end of participation (5 years from baseline at maximum). It will include tumor response and adverse event assessments (AE related to study procedures only)
  Interventions: Other: Tumor biopsy
- Early breast cancer (triple negative, HER2+, luminal) without indication of neo-adjuvant treatment (Other): * The following samples will be collected during the study :
    * Tumor sample (primitive tumor ± metastatic axillary lymph node) at: baseline, surgery, 1st recurrence
    * Blood samples at: baseline (= before surgery), after surgery, end of adjuvant chemotherapy, end of other systemic adjuvant treatment, every 6 or 12 months until the 1st recurrence or during 5 year follow-up period, following progressions/recurrences
    * Ascite and pleural fluid (when a puncture procedure is performed for clinical purposes) at: 1st recurrence, following progressions/recurrences
  * Data collection will be performed at baseline and then at each time point planned in the center for clinical standard of care assessment or clinical trial until end of participation (5 years from baseline at maximum). It will include tumor response and adverse event assessments (AE related to study procedures only)
  Interventions: Other: Tumor biopsy
- De novo metastatic breast cancer (triple negative, HER2+, luminal) (Other): * The following samples will be collected during the study :
    * Tumor sample (primitive tumor ± metastatic axillary lymph node) at: baseline, surgery, 1st progression
    * Blood samples at: baseline, 1st progression, following progressions
    * Ascite and pleural fluid (when a puncture procedure is performed for clinical purposes) at: baseline, 1st progression, following progressions
  * Data collection will be performed at baseline and then at each time point planned in the center for clinical standard of care assessment or clinical trial until end of participation (5 years from baseline at maximum). It will include tumor response and adverse event assessments (AE related to study procedures only)
  Interventions: Other: Tumor biopsy

INTERVENTIONS:
Other: Tumor biopsy — As fresh tumor material is required for laboratory analysis purposes (ESPRESSO technique), tumor biopsies will be performed specifically for this study.

SUMMARY:
This trial is a translational, open-label, monocentric and prospective cohort study of participants with breast cancer aiming to create a combined ESPRESSO (= organelle properties) phenotype and spatial proteomics data collection encompassing four cohorts:

* TN eBC = cohort A,
* HER2+ eBC = cohort B,
* Luminal eBC = cohort C,
* dnMBC = cohort D. In total 1050 participants will be enrolled in the study. Laboratory analysis (including ESPRESSO technique) will be conducted on the biological specimen collected during this study.

The primary objective is to describe the amount of fatty acids accumulated in lipid droplets, within the four cohorts. As a secondary objective, the analysis will expand to other organelles like lysosomal acidity and nuclear organization.

The study is due to last 9 years (4 years of recruitment and 5 years of study participation)

DETAILED DESCRIPTION:
The study targets participants with early breast cancer (eBC) or de novo metastatic breast cancer (dnMBC) who will be treated within a standard of care procedure or a clinical trial.

Following informed consent form signature, participants will be included in the study protocol and will be assigned in one of four cohorts, depending on the immunohistochemical subtype of tumor.

Patients will be enrolled concomitantly in each cohort, with the following recruitment goals:

* Cohort A (N = 300 patients): Triple Negative eBC (TN eBC)
* Cohort B (N = 300 patients): HER2+ eBC (HR+ or HR-)
* Cohort C (N = 300 patients): Luminal eBC (Luminal A or B)
* Cohorte D (N = 150 patients): dnMBC of any subtype (TN, HER2+ or Luminal).

After the cancer treatment completion, the participants will remain in the study for a follow-up period (study participation will be 5 years maximum since baseline).

In this study, anti-cancer procedures or treatments, whatever they are, will not be under investigation; they will be performed, administrated and dosed according to the standard of care or according to the study protocol (if participation in a clinical trial).

For each included participant, biological specimen (fresh tumor sample, blood samples, ascite or pleural fluids if applicable) will be collected. Depending on participant's cohort and treatment strategy (i.e. eBC with indication of neoadjuvant treatment or not, dnMBC with indication of surgical treatment or not), samples will be collected at different times points.

ELIGIBILITY:
* Inclusion Criteria:

  1. Patient (women or men) with histologically documented breast cancer
  2. Early Breast Cancer (eBC) or de novo metastatic BC (dnMBC), regardless the immunohistochemical subtype: Triple Negative BC (ER-negative [<10%], PR-negative [<10%] and HER2-negative [i.e. null, ultra-low or low] BC); HER2-positive BC: HER2 overexpression score 3+ or ERBB2 amplification whatever ER/PR expression and proliferation level; Luminal A-like BC: low to moderately proliferative (Ki67<20%) ER-positive (≥ 10%) PR-positive (≥ 20%) BC and low proliferative (Ki67< 14%) ER-positive PR-negative (< 20%) BC; Luminal B-like BC: highly proliferative (Ki67≥ 20%) ER-positive, PR-positive BC or moderately proliferative (14% ≤ Ki67< 20%) ER-positive PR-negative (<20%) BC
  3. Age ≥ 18 years at the time of study entry
  4. Patient followed within a standard of care procedure or clinical trial
  5. ECOG performance status ≤ 2
  6. Breast cancer treatment not yet started
  7. Patient able to participate and willing to give informed consent prior performance of any study-related procedures and to comply with the study protocol
  8. Patient affiliated to a Social Health Insurance in France.
* Exclusion Criteria:

  1. Known history of positive test for Hepatitis B virus or Hepatitis C virus or Immunodeficiency Virus (HIV) or Hanta virus.
  2. Abnormal coagulation contraindicating biopsy
  3. Previous or on going treatment for the breast cancer
  4. Bone metastases when this is the only site of biopsiable disease for dnMBC patients
  5. Any condition contraindicated with blood sampling procedures required by the protocol (including Hemoglobin < 8g/dl)
  6. Patients with known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
  7. Patient pregnant, or breast-feeding
  8. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure.
  9. Patient who has forfeited his/her freedom by administrative or legal award or who is under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2026-02-06 (Actual); Primary Completion 2035-02-06 (Estimated); Study Completion 2035-02-06 (Estimated)

PRIMARY OUTCOMES:
The amount of fatty acids accumulated in lipid droplets, quantified by the total intensity of a lipid-droplet specific fluorescent dye in the four cohorts | 5 years for each participant

SECONDARY OUTCOMES:
Pathological response will be assessed using residual cancer burden (RCB) index 17 | 5 years for each participant
  * RCB-0: pathologic complete response (pCR)
  * RCB-I : minimal burden
  * RCB-II: moderate burden
  * RCB-III : extensive burden
Event-free survival (EFS) is defined as the time from inclusion until relapse (local, regional or distant) or death from any cause for eBC. | 5 years of each participant
  Participants alive and relapse-free will be censored at last follow-up news or at initiation of new anticancer therapy
First line Progression-free survival (PFS1) is defined as the time from inclusion until progression or death from any cause for dnMBC | 5 years for each participant
  Participants alive and progression-free will be censored at last follow-up news or at initiation of new anticancer therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse, France